CLINICAL TRIAL: NCT06368843
Title: Evaluating the Impact of Ketamine Gargling on Post Intubation Sore Throat: A Randomized Controlled Trial.
Brief Title: the Impact of Ketamine Gargling on the Incidence of Post Intubation Sore Throat
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hussein Ali, lecturer in anesthesiology department, Al-Azhar University
Other Study IDs: Ketamine for POST
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Sore Throat
Keywords: ketamine gargling; Post-operative sore throat; endotracheal tube complications
MeSH Terms: interventions — Mouthwashes; Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- the 1st group (K group): the 1st group (K group) consisted of 46 patients who were instructed to gargle with a ketamine solution
  Interventions: Drug: Gargle with ketamine

INTERVENTIONS:
Drug: Gargle with ketamine — The patients asked to gargling with ketamine solution in the preoperative waiting area after explain the whole procedure and the goals of the study.
  Other Names: Placebo

SUMMARY:
Tracheal intubation often causes trauma to the airway mucosa, leading to postoperative sore throat (POST), which has been reported to occur in 21-65% of cases. While considered a minor complication, POST can contribute to postoperative discomfort and patient dissatisfaction.

DETAILED DESCRIPTION:
Patients have ranked POST as the eighth most adverse effect during the postoperative period. Various methods, both non-pharmacological and pharmacological, have been explored to mitigate POST with varying degrees of success. Non-pharmacological approaches include using smaller-sized endotracheal tubes, lubricating the tube with water-soluble jelly, employing careful airway instrumentation, ensuring intubation after full relaxation, employing gentle oropharyngeal suctioning, minimizing intracuff pressure, and deflating the tracheal tube cuff completely before extubation, all of which have been reported to reduce the incidence of POST.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients from both sex and aged between 18 and 45 years.
* All participants were scheduled for elective laparoscopic appendectomy or cholecystectomy under general anesthesia.
* Classified as ASA (American Society of Anesthesiologists) I or II.
* Intubation duration is less than 90 minutes.

Exclusion Criteria:

* Patients classified as ASA III or higher.
* Patients exhibiting symptoms of sore throat prior to entering the operating room, or presenting with any respiratory illness or signs of respiratory infection.
* Patients who smoke.
* Patients with a history of allergy to drugs used in this study.
* Patients who are addicted to steroid drugs (inhaled or oral).
* Patients with predicted difficult airway and intubation, indicated by a Mallampati score of II or higher.
* Obese patients with a BMI exceeding 35.
* Patients with neurological diseases.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The patients undergoing appendectomy or cholecystectomy under general anesthesia with endotracheal intubation in Al-Nasiriyah Teaching Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Sore throat | 2, 6, 12, and 24 hrs. postoperatively
  A sore throat is characterized by pain, scratchiness, or irritation in the throat, typically aggravated by swallowing.

SECONDARY OUTCOMES:
Cough | 2, 6, 12, and 24 hrs. postoperatively
  Coughing and bucking while intubated on emergence from general anesthesia unfortunately occurs in approximately 40% of patients
Hoarseness of voice | 2, 6, 12, and 24 hrs. postoperatively
  Hoarseness of voice is a common complication after tracheal intubation and may be very limiting for a patient after anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health, Baghdad, Thi-Qar, Iraq

IPD SHARING:
Plan to Share IPD: No
We will not share any data about the participants with other researchers; but we will share the results after doing our analysis.

REFERENCES:
- [Background] Christensen AM, Willemoes-Larsen H, Lundby L, Jakobsen KB. Postoperative throat complaints after tracheal intubation. Br J Anaesth. 1994 Dec;73(6):786-7. doi: 10.1093/bja/73.6.786. PMID 7880666
- [Background] Loeser EA, Bennett GM, Orr DL, Stanley TH. Reduction of postoperative sore throat with new endotracheal tube cuffs. Anesthesiology. 1980 Mar;52(3):257-9. doi: 10.1097/00000542-198003000-00011. No abstract available. PMID 7369513
- [Background] Al-Qahtani AS, Messahel FM. Quality improvement in anesthetic practice--incidence of sore throat after using small tracheal tube. Middle East J Anaesthesiol. 2005 Feb;18(1):179-83. PMID 15830773